CLINICAL TRIAL: NCT03645122
Title: Plasticity in the Spinal Cord to Enhance Motor Retraining After Stroke
Brief Title: Spinal Plasticity to Enhance Motor Retraining After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B2837-W; 1617296 (Other Grant/Funding Number: Veterans Health Administration); NCT03638570 (obsolete NCT alias); NCT03639116 (obsolete NCT alias)
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Cerebrovascular Accident; Hemiparesis
Keywords: Neuromodulation; Transcranial magnetic stimulation (TMS); Electrical stimulation
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: Transcranial magnetic stimulation targeting the region of the brain responsible for voluntary movement control and electrical stimulation to a peripheral nerve innervating hand muscles will be triggered at an interval that elicits action potentials arriving in a set sequence and predetermined delay in the spinal cord.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PCMS REST (Experimental): PCMS will be triggered while the hand/digits are at rest.
  Interventions: Other: Paired corticospinal-motoneuronal stimulation (PCMS)
- SHAM (Active Comparator): SHAM stimulation will be triggered when a criterion level of force stability by the hand/digits is achieved.
  Interventions: Other: Sham stimulation
- PCMS ACTIVE (Experimental): PCMS will be triggered when a criterion level of force stability by the hand/digits is achieved.
  Interventions: Other: Paired corticospinal-motoneuronal stimulation (PCMS)

INTERVENTIONS:
Other: Paired corticospinal-motoneuronal stimulation (PCMS) — Synapses in the spinal cord that transmit voluntary movement commands from the brain to hand muscles will be activated by noninvasive stimulation in a particular sequence and interval that has been shown to strengthen connectivity.
  Arms: PCMS ACTIVE; PCMS REST
Other: Sham stimulation — Synapses in the spinal cord that transmit voluntary movement commands from the brain to hand muscles will not be activated by noninvasive stimulation in a particular sequence and interval that has been shown to strengthen connectivity.
  Arms: SHAM

SUMMARY:
The objective of this project is to study the effects of an emerging noninvasive neuromodulation strategy in human stroke survivors with movement-related disability. Muscle weakness after stroke results from the abnormal interaction between cells in the brain that send commands to control movement and cells in the spinal cord that cause muscles to produce movement. The neuromodulation strategy central to this project has been shown the strengthen the physical connection between both cells, producing a change in movement potential of muscles weakened by stroke.

DETAILED DESCRIPTION:
Stroke is a leading cause of serious long-term disability in the United States with 795,000 individuals suffering a new or recurrent stroke each year. In most cases, disability is associated with incomplete motor recovery of the paretic limb. Full recovery is often not achieved, creating a need for neuromodulation strategies that target the physiological mechanisms impaired by stroke to fully harness the adaptive capacity of the nervous system. The neuromodulation protocol that will be tested in these experiments will target connections between the brain and spinal cord with noninvasive stimulation to enhance movement potential of the hand. Individuals who experienced a single stroke at least 6 months ago may be eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 75 years old
* Diagnosis of first-ever stroke
* Stroke onset of at least six months prior to the time of participation

Exclusion Criteria:

* History of seizure or epilepsy
* Ferromagnetic metallic implants, pacemakers, other implanted devices, or ventilators (for subjects undergoing MRI)
* Pregnant or expecting to become pregnant
* Difficulty maintaining alertness and/or remaining still
* Body weight > 300 lbs due to MRI scanner dimensions (for subjects undergoing MRI)
* Cognitive or language impairments that would interfere with the ability to follow simple instructions, as judged by the investigators
* Diagnosis of movement disorder(s) other than stroke

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Urbin, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539

RESULTS

PARTICIPANT FLOW:
Groups:
- PCMS Rest, Sham, PCMS Active: Participants completed 3 conditions in the following randomized order: PCMS Rest, Sham, PCMS Active
- Sham, PCMS Rest, PCMS Active: Participants completed 3 conditions in the following randomized order: Sham, PCMS Rest, PCMS Active
- PCMS Active, Sham, PCMS Rest: Participants completed 3 conditions in the following randomized order: PCMS Active, Sham, PCMS Rest.
- Sham, PCMS Active, PCMS Rest: Participants completed 3 conditions in the following randomized order: Sham, PCMS Active, PCMS Rest
- PCMS Rest, PCMS Active, Sham: Participants completed 3 conditions in the following randomized order: PCMS Rest, PCMS Active, Sham.
- PCMS Active, PCMS Rest, Sham: Participants completed 3 conditions in the following randomized order: PCMS Active, PCMS Rest, Sham.
Period: Overall Study
Arm/Group | PCMS Rest, Sham, PCMS Active | Sham, PCMS Rest, PCMS Active | PCMS Active, Sham, PCMS Rest | Sham, PCMS Active, PCMS Rest | PCMS Rest, PCMS Active, Sham | PCMS Active, PCMS Rest, Sham
Started | 3 | 3 | 4 | 5 | 4 | 4
Completed | 3 | 3 | 4 | 5 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Condition: 1. Rest PCMS: PCMS was administered with the targeted hand muscles at rest.
  2. Sham: Peripheral nerve stimulation was administered and the stimulating coil discharged when subjects achieved a criterion level of force stability during task repetition. The stimulating coil was rotated to prevent activation of the brain, thus, preventing PCMS.
  3. Active PCMS: PCMS was administered when subjects achieved a criterion level of force stability during task repetition.
Arm/Group | Condition
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Motor Control & Learning
Description: A force tracking task will be performed and a measure of variability about the mean force required by the force to be tracked will be computed.
Time Frame: Measured under each condition, with approximately 2 months required for completion of all conditions.
Measure: Mean (Standard Error); unit: Newton
Groups:
- Rest PCMS: PCMS administered with the targeted hand muscles at rest.
- Sham PCMS: Peripheral nerve stimulation administered and the stimulating coil discharged when subjects achieved a criterion level of force stability during task repetition. Stimulating coil rotated to prevent activation of the brain, thus, preventing PCMS.
- Active PCMS: PCMS administered when subjects achieved a criterion level of force stability during task repetition.
Arm/Group | Rest PCMS | Sham PCMS | Active PCMS
Number analyzed (Participants) | 23 | 23 | 23
Newton | 0.339 (0.141) | 0.359 (0.139) | 0.301 (0.115)

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Rest PCMS: PCMS was administered with the targeted hand muscles at rest.
- Sham PCMS: Peripheral nerve stimulation was administered and the stimulating coil discharged when subjects achieved a criterion level of force stability during task repetition. The stimulating coil was rotated to prevent activation of the brain, thus, preventing PCMS.
- Active PCMS: PCMS was administered when subjects achieved a criterion level of force stability during task repetition.
Arm/Group | Rest PCMS | Sham PCMS | Active PCMS
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT03645122/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT03645122/ICF_001.pdf